CLINICAL TRIAL: NCT00706667
Title: Intravenous Ferric Carboxymaltose (Ferinject®) With or Without Erythropoietin for the Correction of Preoperative Anaemia in Patients Undergoing Orthopaedic Surgery
Brief Title: Intravenous Ferric Carboxymaltose (Ferinject®) With or Without Erythropoietin in Patients Undergoing Orthopaedic Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not being able to recuit sufficient patients due to a lack of complience
Sponsor: University of Zurich (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: StV 07-2008
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Placebo for EPO and for Ferinject ®
  Interventions: Drug: Ferinject ®
- 2 (Active Comparator): Only Ferinject ® , Placebo for EPO
  Interventions: Drug: Ferinject ®
- 3 (Active Comparator): Ferinject ® + EPO
  Interventions: Drug: Ferinject ®

INTERVENTIONS:
Drug: Ferinject ® — iv administration in Arm 1 placebo NaCl 0.9% In arm 2 iv administration of Ferinject ® and subcutaneous NaCl 0.9 % as an EPO placebo In arm 3 iv administration of Ferinject ® and subcutaneous EPO

SUMMARY:
Study Design: Single-centre, block randomised, blinded, controlled, phase IIIb, parallel group pilot study.

Primary Objective:

• To evaluate the effect of the administration of ferric carboxymaltose (Ferinject®) with or without erythropoietin vs. no treatment (standard therapy) on the preoperative anaemia status in patients undergoing orthopaedic surgery

Secondary Objective:

* To gain informations for the design of a possible follow-up study
* To evaluate the effect of the administration of ferric carboxymaltose (Ferinject®) with or without erythropoietin vs. no treatment (standard therapy) on pre- and postoperative Hb levels, iron status, transfusion rate, days until discharge.
* To evaluate the tolerability and safety of Ferinject®

Study Centres:

This is a single centre study

Patients:

A total of 75 completed patients (50 patients in the intravenous iron treatment groups and 25 patients in the no treatment group will be recruited.

DETAILED DESCRIPTION:
TREATMENT:

Patients will be randomised 1:1:1 to one of the following groups:

Group I - Ferinject ® and EPO treatment group 25 patients will be randomised to the Ferinject and EPO treatment group.

For each patient, the cumulative total iron requirement will be calculated using the formula of Ganzoni [Ganzoni et al, 1970]:

Iron deficit [mg] = b.w. [kg]† x (target Hb - actual Hb) [g/L] x 0.24†† + depot iron [mg]

† In patients with a body mass index (BMI = weight [kg] / (height [m] x height [m])) >25, a normalised weight will be used to calculate the iron deficit. Normalised weight [kg] = 25 x height [m] x height [m].

†† Factor 0.24 = 0.0034 (iron content Hb = 0.34%) * 0.07 (blood volume = 7% of b.w.) * 1000 (conversion g to mg) Target Hb: 150 g/L Actual Hb: Value obtained at screening visit Depot iron: 500 mg

Patients will receive a first dose of 1000 mg iron as Ferinject® 21 days prior to the scheduled surgery. Patients will receive Ferinject® once weekly for up to two occasions (Day -21 and Day -14) until the calculated cumulative dose is reached for that individual. The Day -14 infusion may not be necessary, depending on the calculated total iron requirement for each patient. Patients in treatment group 1 will get additionally a single 10000 IU dose of EPO together on treatment day -14.

Group II - Ferinject ® treatment group 25 patients will be randomised to the Ferinject without EPO.

For each patient, the cumulative total iron requirement will be calculated using the formula of Ganzoni [Ganzoni et al, 1970]:

Iron deficit [mg] = b.w. [kg]† x (target Hb - actual Hb) [g/L] x 0.24†† + depot iron [mg]

† In patients with a body mass index (BMI = weight [kg] / (height [m] x height [m])) >25, a normalised weight will be used to calculate the iron deficit. Normalised weight [kg] = 25 x height [m] x height [m].

†† Factor 0.24 = 0.0034 (iron content Hb = 0.34%) * 0.07 (blood volume = 7% of b.w.) *1000 (conversion g to mg) Target Hb: 150 g/L Actual Hb: Value obtained at screening visit Depot iron: 500 mg

Patients will receive a first dose of 1000 mg iron as Ferinject 21 days prior to the scheduled surgery. Patients will receive Ferinject® once weekly for up to two occasions (Day -21 and Day -14) until the calculated cumulative dose is reached for that individual. The Day -14 infusion may not be necessary, depending on the calculated total iron requirement for each patient.

Group III - Control group 25 patients will receive the standard treatment for this patient population (no anaemia treatment).

Primary Efficacy Endpoints

• Hb increase from baseline till day of surgery

Secondary Efficacy Endpoints

* Percentage of patients reaching an Hb of > 12 g/dl (women) or of > 13 g/dl (men) at any point in time during the study
* Change in Hb level from baseline to highest Hb level during the study
* Change in Ferritin value from baseline to highest ferritin value during the study
* Change in Tsat value from baseline to highest Tsat value during the study
* Transfusion rate
* Infection rate
* Days until discharge from hospital
* Days until rehabilitation therapy

Secondary Safety Endpoints:

* Adverse events: type, nature, incidence and outcome
* Vital signs (temperature, blood pressure and heart rate)
* Clinical laboratory panels (haematology/coagulation, clinical chemistry, except Hb and iron status, which are considered to be efficacy endpoints)

Laboratory parameters:

Hematology/coagulation parameters to be analysed are Hb, haematocrit (Hct), red blood cell count (RBC), white blood cell count (WBC) with differential and platelet count, mean corpuscular volume (MCV), mean corpuscular haemoglobin (MCH), mean corpuscular haemoglobin concentration (MCHC).

Clinical chemistry parameters to be analysed are alkaline phosphatase (AP), gamma-glutamyl transpeptidase (GGT), aspartate aminotransferase (AST), alanine aminotransferase (ALT), C-reactive protein (CRP), endogenous erythropoietin.

Iron status parameters include serum iron, serum ferritin, serum transferrin and TSAT.

Additional parameters - folic acid, vitamin B12 and beta-HCG will be analysed at baseline only, creatinin, soluble transferrin receptor and total bilirubin will be analysed at all visits.

Statistical Methods:

Summary statistics will be provided for safety and efficacy parameters as well as for the patients' demographic characteristics. Data will be presented per visit, if appropriate. The test for the primary endpoint is confirmative. Statistical tests of secondary endpoints will be employed for exploratory purposes to highlight interesting comparisons (e.g., baseline versus end of study) that may warrant further consideration. Unless otherwise specified, the significance level of all statistical tests will be 5% with a two-sided alternative. If appropriate, corresponding 95%-confidence intervals will be calculated. The sample size estimation is based on t-test calculation.

Continuous variables will be summarized as mean +/- SD and median with range where appropriate. Continuous variables will be compared using the Kruskal-Wallis test followed by pairwise Mann-Whitney tests with Bonferroni-correction. Nominal variables will be compared using the chi-square test or Fisher's exact test where appropriate. Changes within groups of nominal variables will be analyzed using McNemar test.

Changes within groups of continuous variables will be analyzed using the Friedman test followed by pairwise post hoc comparisons using the Wilcoxon signed rank test with Bonferroni correction. Prevalence of anaemia will be presented with exact confidence interval (CI). Continuous variables will be transformed to normal distribution, and CIs for the mean will be computed. The limits of these CIs then will be retransformed to the original units and interpreted as CIs for the median.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age and signed written informed consent
* Patients scheduled to undergo major orthopaedic surgery (hip or knee arthroplasty or back surgery)
* 10 g/dl < Hb < 13.0 g/dl for men and 10 g/dl < Hb < 12.0 g/dl for women, at screening ( 3 weeks prior to surgery)
* Ferritin < 100 μg/l or 100-300 with TSat < 20%

Exclusion Criteria:

* Suspicion of iron overload (Ferritin >300 μg/l or/and TSAT>50%)
* Active severe infection/inflammation (defined as serum CRP > 20 mg/l) or diagnosed malignancy
* Folate-and/or Vitamin B12 deficiency (according to local lab reference range)
* Known history of hepatitis B/C or HIV-positive
* Liver values 3 times higher than normal
* Immunosuppressive or myelosuppressive therapy
* A concurrent medical condition(s) that, in the view of the investigator, would prevent compliance or participation or jeopardize the health of the patients.
* Pregnancy or lactation
* Transfusion within 1 month prior to study inclusion, EPO treatment with in the last 4 weeks, any iron treatment within 4 weeks prior to the inclusion in the trail
* Participation in any other therapeutic trial within the previous month
* History of thromboembolic events in the family or the patient
* Severe peripheral, coronary or carotid artery disease
* Bodyweight < 50 kg
* Patients not able to understand the German language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Hb increase from baseline till day of surgery | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Theusinger, MD, Principal Investigator — University Hospital Zurich, Division of Anaesthesiology
Locations (1):
- University Hospital Zurich, Division of Anaesthesiology, Zurich, Canton of Zurich, Switzerland